CLINICAL TRIAL: NCT05216159
Title: Effects of a Mobile Health-Health Action Process Approach Based Intervention on Sedentary Behaviour and Stress Among Desk-Basked Office Working Adults
Brief Title: Mobile Health-Health Action Process Approach Based Intervention on Sedentary Behaviour and Stress in Office Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Dr. Harry Prapavessis, Professor, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 120488
Record Dates: First submitted 2022-01-17; First posted 2022-01-31 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Sedentary Behavior; Health Behaviour Change; Perceived Stress
Keywords: Sedentary Behaviour; Health Behaviour Change; Perceived Stress; Health Action Process Approach; Office Workers; mHealth; Mobile Health
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Upon obtaining consent, eligible participants will be randomly assigned to either the intervention group or the control group. The study will run for eight weeks, with a four week intervention period and a follow-up at the end of week eight.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mHealth HAPA Intervention Group (Experimental): This intervention group will receive a single one-on-one behavioural counselling session and weekly action and coping planning worksheets delivered through a downloaded smartphone application with the aim of increasing the breaking of consecutive work related sedentary behaviour. Counselling strategies will be grounded in the HAPA model, specifically focusing on the creation of action plans and the development of coping strategies to increase sedentary behaviour breaks. The weekly HAPA based worksheets will be sent out to participants at the beginning of their work week so that they can formulate their own personal action plans and coping strategies for the week to come. They will be prompted to refer back to the information conveyed in one-on-one counselling session where they should try to create action plans that are specific and meaningful to them. The intervention will last for a total of four weeks with the outcomes being measured through questionnaires.
  Interventions: Behavioral: HAPA behavioural counselling + weekly HAPA worksheets
- Control Group (No Intervention): The control group will receive no intervention or further instruction past the letter of information.

INTERVENTIONS:
Behavioral: HAPA behavioural counselling + weekly HAPA worksheets — Behavioural counselling grounded in the Health Action Process Approach (HAPA; ie., action planning and coping planning) paired with weekly HAPA based worksheets delivered through a mobile application, SEMA3, to reduce consecutive workplace sedentary behaviour.
  Arms: mHealth HAPA Intervention Group

SUMMARY:
This study will explore the effectiveness of a Health Action Process Approach (HAPA) mobile health (mHealth) intervention on reducing sedentary behaviour and perceived stress in desk-based office workers. Half of participants will receive a mHealth HAPA intervention consisting of a theory-driven behavioural counselling session and weekly HAPA based worksheets delivered through a mobile application. The other half of participants will act as a control group and will receive no intervention or information past the letter of information. The study will take place over eight weeks, with the first four weeks acting as the intervention period and a follow-up at the end of week eight.

DETAILED DESCRIPTION:
This two-arm, repeated measure randomized control trial will randomize participants into two groups, an intervention group and a no-contact control group in an attempt to reduce sedentary behaviour in desk-based office workers. The study will last for eight weeks, comprising of a four week intervention period and a follow-up at week eight.

Participants will be full time desk-based office workers primarily recruited from large businesses and corporations. The primary objective of the study is to reduce sedentary behaviour, while the secondary objective is to determine if a theory-based behaviour change intervention tailored to workplace sedentary would affect general stress levels of desk-based office workers over the course of the intervention.

The intervention group will receive an initial theory-based behaviour change counselling session through video chat and then continued through a mobile application where weekly worksheets will be delivered to a participant's mobile phone and encourage the participant to create their own personal and specific action plans and coping strategies. The control group will receive no intervention or further instruction past the letter of information.

Sedentary behaviour will be collected in the form of duration of time spent sitting, frequency of sedentary behaviour breaks, and duration of sedentary behaviour breaks. These variables will be measured through a sedentary behaviour and perceived stress questionnaires that will be delivered through a downloadable mobile phone application.

Outcome measures will be compared within and between groups to detect differences. Participants will be recruited through emails to relevant liaisons and senior executives as well as through emails directly to office working employees in the London area.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* full-time employee in a desk-based office job (work from home accepted)
* have access to a smartphone with internet connection
* can read and write in English

Exclusion Criteria:

* any medical or physical limitation that would prevent standing, stretching, and/or light physical activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Changes in Time Spent Sitting at Work | Baseline, Weeks 1, 2, 3, 4, 8
  modified Occupational Physical Activity Questionnaire (Reis et al., 2005; Chau et al., 2012); 5-items
Changes in Time Spent Standing at Work | Baseline, Weeks 1, 2, 3, 4, 8
  modified Occupational Physical Activity Questionnaire (Reis et al., 2005; Chau et al., 2012); 5-items
Changes in Time Spent Engaged in Light-Intensity Physical Activity at Work | Baseline, Weeks 1, 2, 3, 4, 8
  modified Occupational Physical Activity Questionnaire (Reis et al., 2005; Chau et al., 2012); 5-items
Changes in Frequency of Breaks from Sitting at Work | Baseline, Weeks 1, 2, 3, 4, 8
  Modified version of the Last 7-day Sedentary Behaviour Questionnaire (SIT-Q 7d) (Wijndaele et al., 2014; Sui & Prapavessis, 2016); 1-item; 12-point scale (Less than every 30 min, Every 30-45 min, Every 45 min-1 hour, Every 1-1.5 hours, Every 1.5-2 hours, Every 2-3 hours, Every 3-4 hours, Every 4-5 hours, Over every 5 hours, No interruption); Lower values represent a better outcome
Changes in Duration of Breaks from Sitting at Work | Baseline, Weeks 1, 2, 3, 4, 8
  Modified version of the Last 7-day Sedentary Behaviour Questionnaire (SIT-Q 7d) (Wijndaele et al., 2014; Sui & Prapavessis, 2016); 1-item; 10-point scale (Less than 30 sec, 30 sec-1 min, 1-2 min, 2-3 min, 3-4 min, 4-5 min, 5-10 min, 10-15 min, 15-30 min, Over 30 min); Higher values represent a better outcome

SECONDARY OUTCOMES:
Changes in Perceived Stress | Baseline, Week 4
  Perceived Stress Scale (PSS) (Cohen, Kamarck & Mermelstein, 1983); 10-item; 5-point scale (Never, Almost NEver, Sometimes, Fairly Often, Very Often); Lower values represent a better outcome

OTHER OUTCOMES:
Age | Baseline
  Assessed with a single item question: "What is your age?"
Sex | Baseline
  Assessed with a single item question: "What is your sex?"
Gender | Baseline
  Assessed with a single item question: "What gender do you most identify with?"
Ethnicity | Baseline
  Assessed with a single item question: "What ethnicity do you most identify with?"
Work Environment | Baseline
  Assessed with a three item question: "What is your current work environment?"; in office, at home, hybrid
Type of Occupation | Baseline
  Assessed with a four item question: "What general sector does your occupation fall under?"; private, public, charity, other
Hours of Work per Week | Baseline
  Assessed with a single item question: "What are your typical hours of work on an average week?"
Education Level | Baseline
  Assessed with a single item question: "What is your current formal education level?"

CONTACTS AND LOCATIONS:
Overall Officials: Harry Prapavessis, Ph.D, Principal Investigator — Western University
Locations (1):
- The University of Western Ontario, London, Ontario, Canada